CLINICAL TRIAL: NCT01552018
Title: Saxagliptin and Atherosclerosis. A Possible Role for Saxagliptin in the Prevention of Atherosclerosis Beyond Glucose Metabolism.
Brief Title: Saxagliptin and Atherosclerosis
Acronym: SAXATH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011/773b (REK)
Record Dates: First submitted 2012-02-22; First posted 2012-03-13 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus Type 2
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin (Active Comparator): Saxagliptin 5 mg/day
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — Saxagliptin 5 mg, 1 tablet per day for 3 months
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Placebo — Placebo, 1 tablet per day for 3 months.
  Arms: Placebo

SUMMARY:
Dipeptidyl peptidase 4 (DPP-4) inhibitors are approved as add on therapy to improve glycaemic control in Type 2 Diabetes Mellitus (T2DM). DPP-4 inactivates the incretin hormone glucagon-like peptide 1 (GLP-1). Inhibiting the inactivation of GLP-1 leads to increased insulin- and reduced glucagon secretion after meals. DPP-4 has been shown to be present in atherosclerotic plaques. DPP-4 is a protease with substrates including cytokines and chemokines associated with atherosclerosis/inflammation.

The purpose of this study is to explore the effects of 3 months intervention with DPP-4 inhibitor saxagliptin on biomarkers related to atherosclerosis in patients with stable coronary artery disease (CAD) and T2DM, on circulating levels and on expression levels in circulating monocytes and adipose tissue.

A reduction in markers associated with atherosclerosis could indicate an antiatherosclerotic effect of DPP-4 inhibitors beyond glycaemic control alone.

Due to reduced sample size (recruitment problems) the main focus has changed and will now be on cellular aspects and gene regulation (initially secondary outcome measure).

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18, < 80 years old, with type 2 diabetes mellitus and angiographically proven coronary artery disease.
* HbA1c > 6.5% and under treatment with either metformin and/or glimepiride.

Exclusion Criteria:

* Allergy or hypersensitivity to any of the drug's components.
* Heart failure in NYHA class III or IV.
* Severe liver failure, moderate or severe kidney failure
* Malignant disease.
* Active infectious disease.
* Acute coronary syndrome in the last 3 months.
* Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers | Changes in biomarkers from baseline to 3 months
  A selection of biomarkers associated with atherosclerosis, circulating levels and gene expression levels in adipose tissue and leukocytes.

SECONDARY OUTCOMES:
Gene expression of DPP-4 in adipose tissue and leukocytes | Change in expression level of DPP-4 from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ida U Njerve, MD, Principal Investigator — Center for Clinical Heart Research, Dept. of Cardiology, Oslo University Hospital Ullevaal, Norway
Locations (1):
- Center for Clinical Heart Research, Dept. of Cardiology, Oslo University Hospital Ullevaal, Oslo, Norway